CLINICAL TRIAL: NCT01226966
Title: Conditions for Prescribing Liraglutide in Medical Practice and Assessment of Maintenance Level, Tolerability, and Efficacy of Victoza® (Liraglutide) in Subjects With Type 2 Diabetes
Brief Title: Observational Study on Efficacy and Safety of Liraglutide in Subjects With Type 2 Diabetes
Acronym: EVIDENCE
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN2211-3815; U1111-1116-2722 (Other: WHO)
Record Dates: First submitted 2010-10-20; First posted 2010-10-22 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: liraglutide

INTERVENTIONS:
Drug: liraglutide — Prescription is done at the discretion of the prescribing physician as part of normal clinical routine.

SUMMARY:
This observational study is conducted in Europe. The aim of this non-interventional (observational) study is to evaluate the efficacy of liraglutide (Victoza®) and to assess the conditions of use of Victoza® in daily medical practice in France.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with type 2 diabetes
* Patients having recently started (for less than one week) or starting liraglutide (Victoza®) treatment

Exclusion Criteria:

* Hypersensitivity (allergy) to liraglutide or to any of the excipients
* Patient is participating in a clinical trial at the inclusion
* Type 1 diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients starting or having recently started liraglutide treatment for less than one week, and satisfying the study inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 3152 (Actual)
Dates: Start 2010-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Percentage of patients still in liraglutide treatment and having a HbA1c (glycosylated haemoglobin) value below 7.0% | Month 24

SECONDARY OUTCOMES:
Change in HbA1c at month 3 | Month 0, Month 3
Change in HbA1c at month 6 | Month 0, Month 6
Change in HbA1c at month 12 | Month 0, Month 12
Change in HbA1c at month 18 | Month 0, Month 18
Change in HbA1c at month 24 | Month 0, Month 24
Change in fasting plasma glucose (FPG) at month 3 | Month 0, Month 3
Change in fasting plasma glucose (FPG) at month 6 | Month 0, Month 6
Change in fasting plasma glucose (FPG) at month 12 | Month 0, Month 12
Change in fasting plasma glucose (FPG) at month 18 | Month 0, Month 18
Change in fasting plasma glucose (FPG) at month 24 | Month 0, Month 24
Change in Body Weight at Month 3 | Month 0, Month 3
Change in Body Weight at Month 6 | Month 0, Month 6
Change in Body Weight at Month 12 | Month 0, Month 12
Change in Body Weight at Month 18 | Month 0, Month 18
Change in Body Weight at Month 24 | Month 0, Month 24

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Medical Advisor, Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Paris La Défense Cedex, France

REFERENCES:
- [Result] Gautier JF, Martinez L, Penfornis A, Eschwege E, Charpentier G, Huret B, Madani S, Gourdy P. Effectiveness and Persistence with Liraglutide Among Patients with Type 2 Diabetes in Routine Clinical Practice--EVIDENCE: A Prospective, 2-Year Follow-Up, Observational, Post-Marketing Study. Adv Ther. 2015 Sep;32(9):838-53. doi: 10.1007/s12325-015-0245-x. Epub 2015 Sep 30. PMID 26424330
- [Result] Martinez L, Penfornis A, Gautier JF, Eschwege E, Charpentier G, Bouzidi A, Gourdy P. Effectiveness and Persistence of Liraglutide Treatment Among Patients with Type 2 Diabetes Treated in Primary Care and Specialist Settings: A Subgroup Analysis from the EVIDENCE Study, a Prospective, 2-Year Follow-up, Observational, Post-Marketing Study. Adv Ther. 2017 Mar;34(3):674-685. doi: 10.1007/s12325-017-0476-0. Epub 2017 Jan 30. PMID 28138803
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com